CLINICAL TRIAL: NCT04711564
Title: The Effects of Different Lipid Emulsions on the Adipokines, Inflammatory Markers and Mortality in Critically Ill Patients With Sepsis
Brief Title: The Effects of Different Lipid Emulsions on the Adipokines in Critically Ill Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Collaborators: Turkish Society of Clinical Enteral and Parenteral Nutrition (Other)
Responsible Party: Principal Investigator, Hulya ULUSOY, Clinical Professor, Karadeniz Technical University
Other Study IDs: 23618724
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Sepsis
Keywords: Parenteral Nutrition; Sepsis; Adipokines; Inflammation; Intensive Care
MeSH Terms: conditions — Sepsis; Hyperphagia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipokines (adiponectin, rezistin leptin and visfatin) and cytokines (IL-6, IL-10, IL-1β and TNF-α) in critically ill with sepsis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Provision of olive oil emulsions in PN: Olive oil-based (Oliclinomel: 80% OO, 20% LCT provided in a complete all-in-one PN bag by Baxter) parenteral nutrition
  Interventions: Other: Olive oil-based intravenous fat emulsions
- Provision of soybean emulsions in PN: Soybean-based (Kabiven: 100% LCT provided in a complete all-in-one PN bag)
  Interventions: Other: Soybean-based intravenous fat emulsions

INTERVENTIONS:
Other: Olive oil-based intravenous fat emulsions — Parenteral nutrition planned according to the requirements of the patients is given for ten days.
  Groups: Provision of olive oil emulsions in PN
Other: Soybean-based intravenous fat emulsions — Parenteral nutrition planned according to the requirements of the patients is given for ten days.
  Groups: Provision of soybean emulsions in PN

SUMMARY:
Intravenous lipid emulsions contain a number of biologically active ingredients, but the most important are fatty acids. Different fatty acids can affect a number of different physiological processes in different ways in critically ill patients. Adipose tissue can play an important role in metabolic changes of critical illnesses and in adaptation to stress through structural as well as functional changes Although it is known that serum adipokine and cytokine response changes in critical sepsis patients, the factors affecting these changes and the metabolic consequences of these changes are not well defined. The aim of this study was to evaluate the effects of intravenous lipid emulsions on serum adipokine and cytokine levels in patients with sepsis. Secondly, this is to determine the adipokine and cytokine kinetics in the sepsis process and their relationship with mortality in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sepsis within the last 24 h
* Age above 18 and below 85 years
* Indication of only parenteral nutrition therapy

Exclusion Criteria:

* Planning any different medical nutrition therapy such as enteral nutrition, immunonutrition or oral nutrition
* Hypersensitivity (fish, egg or soy protein)
* Uncontrolled hemorrhage
* Uncontrolled hyperlipidemia
* Severe primary blood coagulation diseases
* Acute pancreatitis
* Acute thromboembolic diseases
* Severe liver failure
* RIFLE stage III and IV renal failure
* Pregnancy or lactation
* Expected stay in ICU not more than 10 days
* Expected survival not more than 10 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis aged 18-85 years given parenteral nutrition therapy
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change of the adipokine in the first ten days in onset sepsis | Baseline and 10 days
  Adipokines levels are assayed using a enzyme-linked immunosorbent assay

SECONDARY OUTCOMES:
Intensive care unit length of stay | Time of admission to the ICU until the time of discharge from the intensive care unit, up to 1 year
  Time from study inclusion to intensive care unit discharge.
28-day mortality | 28 day
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Melda Kangalgil, MSc, Principal Investigator — Karadeniz Technical University; Ahmet Oguzhan Kucuk, MD, Principal Investigator — Karadeniz Technical University; Asiye Ozdemir, MD, Principal Investigator — Karadeniz Technical University; Süleyman Caner Karahan, MD, Principal Investigator — Karadeniz Technical University; Umitcan Ok, MD, Principal Investigator — Karadeniz Technical University; Hatice Bozkurt Yavuz, MD, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University Medical Faculty Department of Anesthesiology and Reanimation, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No